CLINICAL TRIAL: NCT02114060
Title: A Randomized, Double-Blind, Factorial Study to Compare the Safety and Efficacy of Varying Combinations of GEN-003 and Matrix-M2 in Subjects With Genital HSV-2 Infection
Brief Title: Dose Ranging Safety and Efficacy of Therapeutic HSV-2 Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genocea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GEN-003-002
Record Dates: First submitted 2014-04-11; First posted 2014-04-15 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Genital Herpes Simplex Type 2
Keywords: HSV; Herpes; genital infection; vaccine
MeSH Terms: conditions — Herpes Simplex | interventions — Adjuvants, Pharmaceutic; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- GEN-003 Vaccine 30μg / Matrix-M 25μg (Experimental): GEN-003 Vaccine (30 μg of each antigen) with Matrix-M2 adjuvant (25 μg), administered as a 0.5 mL intramuscular (IM) injection.
  Interventions: Biological: GEN-003 Vaccine (30μg of each antigen); Biological: Matrix-M2 Adjuvant (25μg)
- GEN-003 Vaccine 30μg / Matrix-M2 50μg (Experimental): GEN-003 Vaccine (30 μg of each antigen) with Matrix-M2 adjuvant (50 μg), administered as a 0.5 mL intramuscular (IM) injection.
  Interventions: Biological: GEN-003 Vaccine (30μg of each antigen); Biological: Matrix-M2 Adjuvant (50μg)
- GEN-003 Vaccine 30μg / Matrix-M2 75μg (Experimental): GEN-003 Vaccine (30 μg of each antigen) with Matrix-M2 adjuvant (75 μg), administered as a 0.5 mL intramuscular (IM) injection.
  Interventions: Biological: GEN-003 Vaccine (30μg of each antigen); Biological: Matrix-M2 Adjuvant (75μg)
- GEN-003 Vaccine 60μg / Matrix-M2 25μg (Experimental): GEN-003 Vaccine (60 μg of each antigen) with Matrix-M2 adjuvant (25 μg), administered as a 0.5 mL intramuscular (IM) injection.
  Interventions: Biological: GEN-003 Vaccine (60μg of each antigen); Biological: Matrix-M2 Adjuvant (25μg)
- GEN-003 Vaccine 60μg / Matrix-M2 50μg (Experimental): GEN-003 Vaccine (60 μg of each antigen) with Matrix-M2 adjuvant (50 μg), administered as a 0.5 mL intramuscular (IM) injection.
  Interventions: Biological: GEN-003 Vaccine (60μg of each antigen); Biological: Matrix-M2 Adjuvant (50μg)
- GEN-003 Vaccine 60μg / Matrix-M2 75μg (Experimental): GEN-003 Vaccine (60 μg of each antigen) with Matrix-M2 adjuvant (75 μg), administered as a 0.5 mL intramuscular (IM) injection.
  Interventions: Biological: GEN-003 Vaccine (60μg of each antigen); Biological: Matrix-M2 Adjuvant (75μg)
- Placebo (Placebo Comparator): 0.9% Normal Saline administered as a 0.5 mL intramuscular (IM) injection.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GEN-003 Vaccine (30μg of each antigen) — HSV-2 protein subunit vaccine consisting of 2 recombinant T cell antigens: internal fragment of the immediate early (IE) protein ICP and glycoprotein D
  Other Names: HSV Vaccine
  Arms: GEN-003 Vaccine 30μg / Matrix-M 25μg; GEN-003 Vaccine 30μg / Matrix-M2 50μg; GEN-003 Vaccine 30μg / Matrix-M2 75μg
Biological: GEN-003 Vaccine (60μg of each antigen) — HSV-2 protein subunit vaccine consisting of 2 recombinant T cell antigens: internal fragment of the immediate early (IE) protein ICP and glycoprotein D
  Other Names: HSV Vaccine
  Arms: GEN-003 Vaccine 60μg / Matrix-M2 25μg; GEN-003 Vaccine 60μg / Matrix-M2 50μg; GEN-003 Vaccine 60μg / Matrix-M2 75μg
Biological: Matrix-M2 Adjuvant (25μg) — Matrix-M2 is derived from fractionated Quillaja saponins, phosphatidylcholine, and cholesterol.
  Other Names: MM2; Adjuvant
  Arms: GEN-003 Vaccine 30μg / Matrix-M 25μg; GEN-003 Vaccine 60μg / Matrix-M2 25μg
Biological: Matrix-M2 Adjuvant (50μg) — Matrix-M2 is derived from fractionated Quillaja saponins, phosphatidylcholine, and cholesterol.
  Other Names: MM2; Adjuvant
  Arms: GEN-003 Vaccine 30μg / Matrix-M2 50μg; GEN-003 Vaccine 60μg / Matrix-M2 50μg
Biological: Matrix-M2 Adjuvant (75μg) — Matrix-M2 is derived from fractionated Quillaja saponins, phosphatidylcholine, and cholesterol.
  Other Names: MM2; Adjuvant
  Arms: GEN-003 Vaccine 30μg / Matrix-M2 75μg; GEN-003 Vaccine 60μg / Matrix-M2 75μg
Biological: Placebo — 0.9% Normal Saline (NaCl)
  Other Names: 0.9% Normal Saline (NaCl)
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, factorial study to compare the reduction in viral shedding among 6 different combinations of GEN-003, a therapeutic HSV-2 vaccine and Matrix-M2 adjuvant.

Secondary objectives of the study include:

* Evaluation of the safety and tolerability of GEN-003 in combination with Matrix-M2 compared to placebo.
* Comparison of the impact on clinical Herpes Simplex Virus type-2 (HSV-2) disease among the 6 different combinations of GEN-003 antigens and Matrix-M2 adjuvant measured by:

  * Time to first clinical and/or virologic recurrence,
  * Proportion of subjects who are recurrence free at 6 and 12 months after the last dose of vaccine,
  * Lesion rate (percent of days with genital lesions present) during the post-vaccination swabbing periods.
* Evaluation of cellular and humoral responses to GEN-003 antigens.

Additional objectives include:

* Assessment of the correlation between immune responses and change in viral shedding or impact on clinical disease as defined above.
* Determination of the recurrence rate in a subset of subjects not receiving suppressive antivirals throughout the study.

Eligible subjects will enter a baseline period to collect anogenital swabs for 28 consecutive days prior to randomization. Each subject will receive up to 3 doses at 21 day intervals. Subjects will be followed for safety and immunologic response for 12 months following their last dose.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females, ages 18 to 50 years inclusive.
* Diagnosis of genital HSV-2 infection for > 1 year supported by ONE of the following documented in the medical history or performed at screening:

  * Western blot for HSV-2
  * Type-specific polymerase chain reaction (PCR) or viral culture
  * Compatible clinical history AND
* Positive HerpeSelect® 2 Enzyme-linked Immunosorbent Assay (ELISA) Immunoglobulin G (IgG) with an index value >3.5, or
* Positive LIAISON® HSV-2 Type-Specific IgG
* A history of at least 3 and no more than 9 reported clinical occurrences in the prior 12 months, or, if currently on suppressive therapy, history of at least 3 and no more than 9 reported clinical occurrences in the 12 months prior to initiation of suppressive therapy.
* Collection of at least 45 of 56 anogenital swabs during the baseline period.
* Willing and able to provide written informed consent.
* Willing to perform and comply with all study procedures including attending clinic visits as scheduled.
* Men and women of childbearing potential, must be willing to practice a highly effective method of contraception that may include, but is not limited to, abstinence, monogamous relationship with vasectomized partner, vasectomy, licensed hormonal methods, intrauterine device (IUD), or barrier method (e.g., condom, diaphragm) for 28 days before and 90 days after receiving Study Drug.

Exclusion Criteria:

* On suppressive antiviral medication within 7 days of beginning baseline anogenital swab collection period.
* History of genital Herpes Simplex Virus type-1 (HSV-1) infection.
* History of any form of ocular Herpes Simplex Virus (HSV) infection, HSV-related erythema multiforme, or herpes meningitis or encephalitis.
* Immunocompromised individuals, including those receiving immunosuppressive doses of corticosteroids (more than 20 mg of prednisone given daily or on alternative days for 2 weeks or more within 6 months prior to the first dose of Study Drug, any dose of corticosteroids within 30 days of the first dose of Study Drug, or high dose inhaled corticosteroids [> 960 μg/day of beclomethasone dipropionate or equivalent]) or other immunosuppressive agents.
* Presence or history of autoimmune disease, regardless of current treatment.
* Positive serologic test for Human Immunodeficiency Virus (HIV-1) or hepatitis C infection; positive hepatitis B surface antigen (HBsAg).
* Clinically significant laboratory abnormality or a value ≥ Grade 2.
* Prior immunization with a vaccine containing HSV-2 antigens.
* History of hypersensitivity to any component of the vaccine.
* Receipt of any investigational drug within 30 days prior to the first dose of Study Drug.
* Receipt of blood products within 90 days prior to the first dose of Study Drug.
* Receipt of a live vaccine within 28 days prior to or a subunit vaccine within 14 days prior to the first dose of Study Drug or planned vaccination within 30 days following the last dose of Study Drug.
* Pregnant or nursing women.
* History of drug or alcohol abuse that, in the opinion of the Investigator, would interfere with the patient's ability to comply with the requirements of the study.
* Other active, uncontrolled co-morbidities that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with the study requirements.

NOTE: Subjects who are taking a medication to control an underlying co-morbidity may be enrolled if there have been no changes to their medication within 60 days prior to the first dose of Study Drug.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 310 (Actual)
Dates: Start 2014-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in proportion of days with detectable viral shedding | 6 weeks

SECONDARY OUTCOMES:
Immunogenicity measured by humoral (antibody) and T-cell responses to vaccine antigens | 33 weeks
Impact on clinical HSV-2 disease based on time to recurrence and lesion rate | 53 weeks
Number of patients with adverse events as a measure of safety and tolerability | 57 weeks

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - University of Alabama Vaccine Research Unit, Birmingham, Alabama
  - Medical Center for Clinical Research, San Diego, California
  - Quest Clinical Research, San Francisco, California
  - University of Illinois Department of Medicine, Chicago, Illinois
  - Indiana University Infectious Disease Research, Indianapolis, Indiana
  - The Fenway Institute, Boston, Massachusetts
  - UNC Global HIV Prevention and Treatment Clinical Trials Unit, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Westover Heights Clinic, Portland, Oregon
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Tekton Research, Austin, Texas
  - Center for Clinical Studies - Houston, Houston, Texas
  - Center for Clinical Studies, Houston, Texas
  - Center for Clinical Studies - Clear Lake/Webster, Webster, Texas
  - University of Utah, Salt Lake City, Utah
  - UW Virology Research Clinic, Seattle, Washington